CLINICAL TRIAL: NCT06548828
Title: Effects of a Non-nutritive Sweetener Reduction Intervention in Pregnancy and Lactation on Maternal and Infant Outcomes (the SweetPea Trial)
Brief Title: Effects of a Non-nutritive Sweetener Reduction Intervention in Pregnancy and Lactation on Maternal and Infant Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Children's Hospital Los Angeles (Other); Children's National Research Institute (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Allison Sylvetsky (Meni), Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SweetPea; R01HD107427 (NIH)
Record Dates: First submitted 2024-05-01; First posted 2024-08-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Glucose Intolerance During Pregnancy; Non-nutritive Sweeteners Consumption in Pregnancy and/or Lactation
Keywords: Non-nutritive sweeteners (NNS); Pregnancy; Lactation; Infant fat mass; Gestational diabetes (GDM); Glucose tolerance; PeaPod
MeSH Terms: conditions — Breast Feeding; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff will be instructed to assign allocated numbers to participants in sequential order as they are enrolled. Once the assignment (1, 2 or 3) is revealed to the study team, study information per that assignment will be explained to the participant. It is essential for the research team to know the allocation in order to provide the correct intervention materials and relevant counseling. Thus, the design is open-label, with only outcome assessors blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Group 1) (Active Comparator): Participants in this arm will continue their usual consumption of NNS throughout pregnancy and lactation without any intervention. They will not receive any specific NNS-restriction intervention.
  Interventions: Behavioral: Control Intervention
- NNS Restriction in Lactation (Group 2) (Active Comparator): Participants in this arm will maintain their usual NNS consumption during pregnancy but will receive an intervention to restrict NNS intake during lactation.
  Interventions: Behavioral: NNS Restriction Intervention; Behavioral: Control Intervention
- NNS Restriction in Pregnancy and Lactation (Group 3) (Active Comparator): Participants in this arm will receive an intervention to restrict NNS intake both during pregnancy and lactation.
  Interventions: Behavioral: NNS Restriction Intervention

INTERVENTIONS:
Behavioral: NNS Restriction Intervention — Discuss current scientific literature surrounding NNS consumption, obesity, and chronic disease and the emerging evidence that consumption in pregnancy/lactation may have unfavorable effects on infants' adiposity and health.
  Provide detailed handouts, which will include a list of specific foods and beverages containing NNS to avoid during the study and summarize current scientific evidence on the metabolic and health effects of NNS.
  Emphasize that sugar is not the best alternative to NNS, and that the participant should drink still water, sparkling water, flavored waters with no added sweeteners, or unsweetened tea instead.
  Bi-weekly shipments of unsweetened beverages of participant's choice to replace usual consumption of NNS containing beverages.
  Automated text messages will also be sent to mothers once per week with reminders that they should avoid NNS
  Arms: NNS Restriction in Lactation (Group 2); NNS Restriction in Pregnancy and Lactation (Group 3)
Behavioral: Control Intervention — Counsel about best practices for home safety and babyproofing.
  Provide a detailed booklet to take home, which will provide information about home safety and baby proofing.
  Educate about common causes of accidental infant and young child injuries or death.
  Automated text messages will also be sent to mothers once per week with reminders about home safety, infant safety, and baby proofing.
  Arms: Control (Group 1); NNS Restriction in Lactation (Group 2)

SUMMARY:
The effects of consuming non-nutritive sweeteners (NNS) during pregnancy and lactation on infant obesity and cardiometabolic disease risk are not well understood. In this project, pregnant women who frequently consume NNS will be randomly assigned to an NNS-restriction intervention (NNS restriction during pregnancy and lactation or during lactation only) or a control group (no NNS restriction) to determine whether NNS consumption during pregnancy and/or lactation affects infant body composition, maternal blood sugar during pregnancy, and the infants' gut microbiome and metabolome. The results of this study have the potential to shape recommendations around NNS consumption during pregnancy and lactation, thereby potentially improving maternal and infant metabolic health and reducing the global burden of obesity and cardiometabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* ≤ 16 weeks gestation
* Singleton pregnancy
* Report frequent NNS beverage consumption (≥ 7 servings/week)
* 18-45 years of age
* Able to read English at a 5th grade level; and
* Intend to breastfeed for at least the first 6 months of life.
* For infants: The mother must be enrolled and provide assent for the infant to participate.

Exclusion Criteria:

* Physical or mental concerns preventing study participation;
* Medication (e.g., metformin; GLP-1 agonists) use that may affect body weight, body composition, insulin resistance, or lipid profiles;
* Tobacco or drug use during pregnancy;
* Alcohol consumption (>1 drink per week) during pregnancy;
* Pre-existing gastrointestinal, inflammatory, or malabsorptive disorders (e.g., - Crohn's disease, ulcerative colitis, inflammatory bowel disease) that may impact NNS absorption or gut microbiota;
* Known suspected/confirmed genetic fetal abnormalities or suspected or known congenital birth defects.
* History of prior gastric bypass surgery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Infants' adiposity | At 6 months of age
  Determine the impact of restricting usual consumption of non-nutritive sweeteners (NNS) during pregnancy and/or lactation influences infants' adiposity, which is known to be predictive of potential future obesity risk by assess infants' fat mass percent.
Mothers' incremental area under glucose response curves | At 28 weeks gestation
  Determine the impact of restricting usual consumption of non-nutritive sweeteners (NNS) during pregnancy on maternal glucose tolerance by assessing the incremental area under the 120 minute glucose response curves.

SECONDARY OUTCOMES:
Infants' adiposity | At 1 month of age
  Determine the impact of restricting usual consumption of non-nutritive sweeteners (NNS) during pregnancy and/or lactation influences infants' adiposity, which is known to be predictive of potential future obesity risk by assess infants' fat mass percent.
Mothers' fasting blood glucose concentration | At 28 weeks gestation
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy on mothers' metabolic and inflammatory biomarkers by assessing fasting glucose concentrations.
Mothers' fasting blood glucose concentration | At 1 month postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy on mothers' metabolic and inflammatory biomarkers by assessing fasting glucose concentrations.
Mothers' fasting blood glucose concentration | At 6 months postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy on mothers' metabolic and inflammatory biomarkers by assessing fasting glucose concentrations.
Mothers' 60 minute glucose concentration | At 28 weeks gestation
  Determine the impact of restricting usual consumption of non-nutritive sweeteners (NNS) during pregnancy on maternal glucose tolerance by assessing the blood glucose levels 60 minutes following ingestion of a standard glucose/water mixture
Mothers' 120 minute glucose concentration | At 28 weeks gestation
  Determine the impact of restricting usual consumption of non-nutritive sweeteners (NNS) during pregnancy on maternal glucose tolerance by assessing the blood glucose levels 120 minutes following ingestion of a standard glucose/water mixture.
Infants' gestational age | At birth
  Determine gestational age at birth.
Infants' birthweight | At birth
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy and/or lactation on infants' growth by assessing birth weight.
Infants' birthweight based on gestational age | At birth
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy and/or lactation on infants' growth by assessing birth weight for gestational age.
Infants' age-sex specific percentile | At 1 month of age
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy and/or lactation on infants' height and weight for age by assessing age-sex specific percentile.
Infants' age-sex specific percentile | At 6 months of age
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy and/or lactation on infants' height and weight for age by assessing age-sex specific percentile.
Mothers' insulin sensitivity index | At 28 weeks gestation
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy on maternal insulin sensitivity by assessing composite whole-body insulin sensitivity index (WBISI).
Mothers' assessment of insulin resistance | At 28 weeks gestation
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy on maternal insulin sensitivity by assessing homeostasis model assessment of insulin resistance (HOMA-IR).
Mothers' energy intake | At 28 weeks gestation
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during lactation on mothers' mean energy intake from dietary recalls during pregnancy.
Mothers' energy intake | At 1 month postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during lactation on mothers' mean energy intake from dietary recalls during postpartum.
Mothers' energy intake | At 6 months postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during lactation on mothers' mean energy intake from dietary recalls during postpartum.

OTHER OUTCOMES:
Infants' gut microbiome composition | At 1 month of age
  Determine the effects of restricting usual consumption of non-nutritive sweeteners (NNS) during pregnancy and/or lactation on the composition of the infant gut microbiome as it changes dramatically over the first few years of life by evaluating relative abundance of Firmicutes, Akkermansia muciniphila, Bifidobacterium, Lactobacillus, Proteobacteria present in stool specimens.
Infants' gut microbiome composition | At 6 months of age
  Determine the effects of restricting usual consumption of non-nutritive sweeteners (NNS) during pregnancy and/or lactation on the composition of the infant gut microbiome as it changes dramatically over the first few years of life by evaluating relative abundance of Firmicutes, Akkermansia muciniphila, Bifidobacterium, Lactobacillus, Proteobacteria present in stool specimens.
Mothers' gestational weight gain | At delivery
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy on mothers' total weight gain during pregnancy by assessing maternal gestational weight gain (GWG).
Mothers' waist circumference | At 1 month postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during lactation on mothers' adiposity by assessing waist circumference (WC).
Mothers' waist circumference | At 6 months postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during lactation on mothers' adiposity by assessing waist circumference (WC).
Mothers' body composition during pregnancy | At 28 weeks gestation
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy on mothers' body composition by assessing percent body fat.
Mothers' C-reactive protein (CRP) concentration | At 28 weeks gestation
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy and postpartum on mothers' fasting concentration of C-reactive protein (CRP) concentrations.
Mothers' C-reactive protein (CRP) concentration | At 1 month postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy and postpartum on mothers' fasting concentration of C-reactive protein (CRP) concentrations.
Mothers' C-reactive protein (CRP) concentration | At 6 months postpartum
  Determine effects of restricting usual non-nutritive sweeteners (NNS) consumption during pregnancy and postpartum on mothers' fasting concentration of C-reactive protein (CRP) concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States